CLINICAL TRIAL: NCT00494299
Title: Phase III Study of BAY43-9006 in Patients With Advanced Hepatocellular Carcinoma (HCC) Treated After Transcatheter Arterial Chemoembolization (TACE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11721
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Results first posted 2011-01-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; Cancer; Liver Cancer; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib (Nexavar, BAY43-9006) administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid) (morning and evening, every 12 hours as far as possible); Dose modification (delayed or reduced) was permitted due to toxicity.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)
- Placebo (Placebo Comparator): Sorafenib (Nexavar, BAY43-9006) matching placebo (2 placebo tablets) orally administered bid (twice daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Multikinase Inhibitor; Sorafenib: 400mg bid of sorafenib
  Arms: Sorafenib (Nexavar, BAY43-9006)
Drug: Placebo — Placebo: matching placebo
  Arms: Placebo

SUMMARY:
Clinical trial of BAY43-9006 in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged of 18 and over
* Advanced hepatocellular carcinoma

Exclusion Criteria:

* History of prior systemic chemotherapy
* Failure in vital organ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (56):
- Japan (52):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Tōon, Ehime
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Iizuka, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Gifu, Gifu
  - Isesaki, Gunma
  - Maebashi, Gunma
  - Hiroshima, Hiroshima
  - Kure, Hiroshima
  - Sapporo, Hokkaido
  - Akashi, Hyōgo
  - Kobe, Hyōgo
  - Kasama, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Kagoshima, Kagoshima-ken
  - Isehara, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Miyazaki, Miyazaki
  - Matsumoto, Nagano
  - Ōmura, Nagasaki
  - Okayama, Okayama-ken
  - Kawachi-Nagano, Osaka
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Izunokuni, Shizuoka
  - Sunto, Shizuoka
  - Shimotsuke, Tochigi
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Nerima-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Yonago, Tottori
  - Toyama, Toyama
  - Yamagata, Yamagata
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi
  - Chūō, Yamanashi
- South Korea (4):
  - Seoul, Seoul Teugbyeolsi
  - Daegu
  - Incheon
  - Seoul

REFERENCES:
- [Result] Kudo M, Imanaka K, Chida N, Nakachi K, Tak WY, Takayama T, Yoon JH, Hori T, Kumada H, Hayashi N, Kaneko S, Tsubouchi H, Suh DJ, Furuse J, Okusaka T, Tanaka K, Matsui O, Wada M, Yamaguchi I, Ohya T, Meinhardt G, Okita K. Phase III study of sorafenib after transarterial chemoembolisation in Japanese and Korean patients with unresectable hepatocellular carcinoma. Eur J Cancer. 2011 Sep;47(14):2117-27. doi: 10.1016/j.ejca.2011.05.007. PMID 21664811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 27 Aug 2006. The final data collection date for the primary endpoint analysis was 10 Jul 2009. The study was conducted at 77 centers from 2 countries: Korea (7 centers) and Japan (70). 76 centers enrolled at least 1 subject (7 centers in Korea and 69 in Japan). The last subject's last visit occurred on 19 Nov 2010.
Pre-assignment Details: Of 552 subjects screened, 458 were randomized and were valid for the efficacy analyses (intent to treat [ITT] population), and 456 received at least 1 dose of study drug and were valid for the safety analyses. 229 subjects were randomized to each group (sorafenib or placebo).
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Started | 229 | 229
Received Treatment | 229 | 227
Completed | 0 | 0
Not Completed | 229 | 229
Not completed — Adverse Event | 93 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Disease Progression, Recurrence/Relapse | 109 | 185
Not completed — Participant Did Not Take Study Drug | 0 | 2
Not completed — Site Closed by Sponsor | 6 | 0
Not completed — Protocol Driven Decision Point | 11 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo | Total
Number analyzed (Participants) | 229 | 229 | 458
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (8.7) | 68.1 (8.8) | 67.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 61 | 116
  Male | 174 | 168 | 342
Child Pugh Status [Number; unit: Participants] — A Child-Pugh (CP) score (determined by encephalopathy grade, ascites, serum bilirubin and albumin, prothrombin time) is used to assess the prognosis of chronic liver disease, mainly cirrhosis. One of the inclusion criterion for this study was a CP class A (good operative risk); class B (moderate risk) score or class C (poor operative risk) was excluded.
  Participants
    Status A | 229 | 229 | 458
    Status B | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects a patient. 0 = fully active, 1 = restricted strenuous activity, 2 = ambulatory, 3 = limited selfcare, 4 = completely disabled, 5 = dead. Subjects entering this study must have had an ECOG score of 0 or 1.
  Participants
    Grade 0 | 201 | 202 | 403
    Grade 1 | 28 | 27 | 55
    Grade 2 | 0 | 0 | 0
    Grade 3 | 0 | 0 | 0
    Grade 4 | 0 | 0 | 0
Responder group to transcatheter arterial chemoembolization (TACE) [Number; unit: Participants] — Responder Group A: percentage of tumor necrosis or tumor shrinkage is 100 percentage. Responder Group B: percentage of tumor necrosis or tumor shrinkage is 25 percentage or more to less than 100 percentage. Subjects entering this study is a responder to TACE.
  Participants
    Responder Group A | 142 | 142 | 284
    Responder Group B | 87 | 87 | 174
Number of Prior transcatheter arterial chemoembolization (TACE) [Number; unit: Participants] — Subjects entering this study must have had previous TACE at a maximum of 2 times.
  Participants
    1 | 147 | 148 | 295
    2 | 82 | 81 | 163

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from date of randomization to radiological progression / recurrence. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From randomization of the first subject until radiological progression or recurrence whichever came first, assessed up to 39 months.
Population: Intention to treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 229 | 229
days | 164 [116 to 220] | 112 [106 to 122]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Log Rank = 0.25204620 — The comparison between the 2 groups is done using the log rank test stratified by the response of TACE (Responder group A versus Responder group B), ECOG performance status (PS) (0 versus 1) and the number of prior TACE (1 versus 2)
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8735, 95% CI [0.6972 to 1.0942] — Hazard Ratio: Sorafenib/Placebo

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from date of randomization to death due to any cause. Subjects still alive at their last date of follow-up were censored at the time of analysis.
Time Frame: From randomization of the first subject until 39 months later.
Population: Median overall survival (OS) and 95% Confidence interval (CI) were not estimable in Placebo Group and Upper Limit of 95% CI was not in Sorafenib Group because of more than half (188 for Placebo,186 for Sorafenib) of the individual study populations censored. Number of death is shown in "Post-Hoc Outcome Measure".
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 0 | 0

3. Post Hoc Outcome: Number of Death Cases Due to Any Cause
Time Frame: From randomization of the first subject until death due to any cause assessed up to 55 months.
Population: Intention to treat (ITT) population. "Overall Survival" is shown in "Secondary Outcome Measure: Overall Survival".
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Number analyzed (Participants) | 229 | 229
Participants
  up to 39 months | 43 | 41
  up to 55 months | 50 | 56

ADVERSE EVENTS:
Description: Acronyms in Adverse Event section: - Absolute Neutrophil Count (ANC) - Alanine Transaminase (ALT) - Aspartate Transaminase (AST) - Atrioventricular (AV) - Central Nervous System (CNS) - Gastrointestinal (GI) - International Normalized Ratio (INR) - Not Otherwise Specified (NOS)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) | Placebo
Serious Adverse Events (participants affected / at risk) | 44/229 | 21/227
Other Adverse Events (participants affected / at risk) | 229/229 | 193/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=229) | Placebo (N=227)
NEUTROPHILS (Blood and lymphatic system disorders) | 1 | 0
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 | 0
PLATELETS (Blood and lymphatic system disorders) | 1 | 0
INR (Blood and lymphatic system disorders) | 1 | 0
EDEMA: LIMB (Blood and lymphatic system disorders) | 1 | 0
CONDUCTION ABNORMALITY, AV BLOCK-3RD DEGREE (COMPLETE AV BLOCK) (Cardiac disorders) | 0 | 1
CARDIAC ISCHEMIA/INFARCTION (Cardiac disorders) | 2 | 0
DIABETES (Endocrine disorders) | 1 | 0
HYPERTHYROIDISM (Endocrine disorders) | 0 | 1
ANOREXIA (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 4 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DEHYDRATION (Gastrointestinal disorders) | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 3 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
GI - OTHER (SPECIFY) (Gastrointestinal disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1
FEVER (General disorders) | 2 | 0
FATIGUE (General disorders) | 0 | 1
PAIN, BACK (General disorders) | 0 | 1
PAIN, ABDOMEN NOS (General disorders) | 2 | 3
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1
LIVER DYSFUNCTION (Hepatobiliary disorders) | 1 | 0
HEPATOBILIARY - OTHER (SPECIFY) (Hepatobiliary disorders) | 3 | 0
INFECTION (DOCUMENTED CLINICALLY), LUNG (PNEUMONIA) (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, BLOOD (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, BILIARY TREE (Infections and infestations) | 2 | 0
INFECTION WITH NORMAL ANC, LIVER (Infections and infestations) | 1 | 0
INFECTION WITH NORMAL ANC, LUNG (PNEUMONIA) (Infections and infestations) | 2 | 0
INFECTION WITH NORMAL ANC, SKIN (CELLULITIS) (Infections and infestations) | 0 | 1
ALT (Metabolism and nutrition disorders) | 2 | 0
AMYLASE (Metabolism and nutrition disorders) | 1 | 0
AST (Metabolism and nutrition disorders) | 2 | 0
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 3 | 0
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0
LIPASE (Metabolism and nutrition disorders) | 1 | 0
METABOLIC/LAB - OTHER (SPECIFY) (Metabolism and nutrition disorders) | 4 | 1
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL - OTHER (SPECIFY) (Musculoskeletal and connective tissue disorders) | 1 | 1
CNS ISCHEMIA (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 6 | 2
MOOD ALTERATION, DEPRESSION (Nervous system disorders) | 1 | 0
SYNCOPE (FAINTING) (Nervous system disorders) | 0 | 1
RENAL - OTHER (SPECIFY) (Renal and urinary disorders) | 0 | 2
HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 3 | 0
DERMATOLOGY - OTHER (SPECIFY) (Skin and subcutaneous tissue disorders) | 0 | 1
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 | 0
CNS HEMORRHAGE (Vascular disorders) | 3 | 0
HEMORRHAGE, GI, ABDOMEN NOS (Vascular disorders) | 0 | 1
HEMORRHAGE, GI, COLON (Vascular disorders) | 0 | 1
HEMORRHAGE, GI, ESOPHAGUS (Vascular disorders) | 1 | 0
HEMORRHAGE, GI, VARICES (ESOPHAGEAL) (Vascular disorders) | 2 | 1
HEMORRHAGE, GI, STOMACH (Vascular disorders) | 1 | 0
HEMORRHAGE, GI, LIVER (Vascular disorders) | 0 | 1
HEMORRHAGE, GI, LOWER GI NOS (Vascular disorders) | 1 | 0
ARTERY INJURY, AORTA (Vascular disorders) | 1 | 0
VASCULAR - OTHER (SPECIFY) (Vascular disorders) | 2 | 0
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=229) | Placebo (N=227)
NEUTROPHILS (Blood and lymphatic system disorders) | 35 | 16
LYMPHOPENIA (Blood and lymphatic system disorders) | 17 | 8
PLATELETS (Blood and lymphatic system disorders) | 64 | 10
LEUKOCYTES (Blood and lymphatic system disorders) | 23 | 15
EDEMA: LIMB (Blood and lymphatic system disorders) | 30 | 20
HYPERTENSION (Cardiac disorders) | 76 | 21
ANOREXIA (Gastrointestinal disorders) | 45 | 18
ASCITES (Gastrointestinal disorders) | 27 | 10
CONSTIPATION (Gastrointestinal disorders) | 30 | 21
DIARRHEA (Gastrointestinal disorders) | 81 | 27
DISTENSION (Gastrointestinal disorders) | 13 | 4
HEARTBURN (Gastrointestinal disorders) | 15 | 16
MUCOSITIS (FUNCTIONAL/SYMPTOMATIC), ORAL CAVITY (Gastrointestinal disorders) | 26 | 5
MUCOSITIS (CLINICAL EXAM), ORAL CAVITY (Gastrointestinal disorders) | 13 | 6
NAUSEA (Gastrointestinal disorders) | 26 | 18
VOMITING (Gastrointestinal disorders) | 16 | 11
FEVER (General disorders) | 37 | 25
WEIGHT GAIN (General disorders) | 4 | 12
FATIGUE (General disorders) | 46 | 34
WEIGHT LOSS (General disorders) | 28 | 3
PAIN, BACK (General disorders) | 13 | 19
PAIN, EXTREMITY-LIMB (General disorders) | 12 | 11
PAIN, ABDOMEN NOS (General disorders) | 29 | 21
PAIN, HEAD/HEADACHE (General disorders) | 25 | 21
PAIN, JOINT (General disorders) | 10 | 15
FLU-LIKE SYNDROME (General disorders) | 44 | 56
INFECTION - OTHER (SPECIFY) (Infections and infestations) | 12 | 6
ALKALINE PHOSPHATASE (Metabolism and nutrition disorders) | 16 | 5
ALT (Metabolism and nutrition disorders) | 59 | 29
AMYLASE (Metabolism and nutrition disorders) | 51 | 18
AST (Metabolism and nutrition disorders) | 70 | 29
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 36 | 12
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 12 | 11
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 19 | 5
LIPASE (Metabolism and nutrition disorders) | 105 | 19
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 79 | 22
METABOLIC/LAB - OTHER (SPECIFY) (Metabolism and nutrition disorders) | 86 | 27
PROTEINURIA (Metabolism and nutrition disorders) | 31 | 1
MUSCULOSKELETAL - OTHER (SPECIFY) (Musculoskeletal and connective tissue disorders) | 19 | 12
NEUROPATHY: SENSORY (Nervous system disorders) | 13 | 9
VOICE CHANGES (Respiratory, thoracic and mediastinal disorders) | 35 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 95 | 8
HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 188 | 17
DERMATOLOGY - OTHER (SPECIFY) (Skin and subcutaneous tissue disorders) | 13 | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 26 | 31
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 99 | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less